CLINICAL TRIAL: NCT04855318
Title: The Effect of Plethysmographic Variability Index Monitoring on Fluid Replacement in Bariatric Surgery
Brief Title: Fluid Replacement in Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, assistant professor, Marmara University
Other Study IDs: 09.2020.158
Record Dates: First submitted 2021-04-04; First posted 2021-04-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: obesity; fluid therapy; pleth variability index
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The frequency of obese postoperative rhabdomyolized acute tubular necrosis (ATN) and renal failure is also increasing. It is simply important to manage fluid. The fluid requirement should be higher than planned. In order to learn the postoperative ATN and the development of renal failure, 4-5 lt crystalloid fluid should be given in 2-3 times or 1.5 ml / kg / h should be provided in the upper outlet.

According to TVA, there are no good guidelines for intraoperative fluid management in bariatric surgery. Different intraoperative fluid management communications are used. The key to improving outcomes from post-operative treatment is "patient directed fluid management" or "targeted fluid management". The use of Perioperative Goal-Directed Fluid Therapy Technologies helps the anesthesiologist closely monitor the patient and strike the delicate balance between benefit and risk. Plethysmographic variability index monitoring (PVI-Pleth Variability Index) is a non-invasive, automatic and continuous monitor that displays patient fluid response, it is one of the easily applicable and easily interpreted monitoring methods. With PVI monitoring, intraoperative hypotension and fluid need can be predicted in advance.

Plethysmographic Variability Index (PVI) is the determination of the importance of monitoring of intraoperative volume replacement and its effect on postoperative operations.

DETAILED DESCRIPTION:
Obesity is defined as an increase in body weight beyond requirements as a result of excessive fat accumulation in the body and is common Obesity leads to an increase in health problems and morbidity and mortality, as well as individual and social problems and a decrease in the workforce. Despite sports, diet, lifestyle changes and medical treatments, the rate of obesity continues to increase in the population. The most effective and durable treatment option for morbid obesity is bariatric surgery. Video laparoscopic bariatric surgery (VLBS) is recognized as the best surgical technique for morbidly obese individuals with health complications associated with excess body fat. Despite the proven benefits of VLBS, it can model a systemic inflammatory response. VLBS also poses an inherent risk of pneumoperitoneum for the kidneys due to high intra-abdominal pressure, which reduces cortical capillary blood flow by increasing renal vascular resistance. As a result, the glomerular filtration rate (GFR) decreases and transient oliguria occurs. Acute renal failure manifested as a large increase in creatinine levels with oliguria.

It is a preventable complication with intraoperative anesthesia management.Glomerular filtration rate (GFR) and increased renal plasma flow cause hyperfiltration syndrome in obesity. Adinopectin, proinflammatory cytokines, oxidative stress and pharmacological nephrotoxicity are the mechanisms affecting acute kidney injury in obesity. Chronic renal failure occurs as a result of a decrease in albiminuria and GFR. They are the causes of postoperative renal failure in patients with diabetes, a history of kidney disease, using antihypertensive drugs containing diuretics, and obese patients with a BMI greater than 50 kg / m2, prolonged operation time, and intraoperative hypotension.

The frequency of acute tubular necrosis (ATN) and renal failure due to postoperative rhabdomyolysis is also increased in obese patients. Fluid management is important to prevent this. The fluid requirement should be higher than planned. In order to prevent the development of postoperative ATN and renal failure, 4-5 liters of crystalloid fluid should be given in 2-3 hours or urine output above 1.5 ml / kg / h should be provided.

According to TVA, there are studies performing crystalloid fluid replacement in a wide range of 15-40 ml / kg.

In obese patients, changes in distribution volume such as decreased hepatic blood flow, increase in renal blood flow and glomerular filtration rate and increase in the amount of free-flowing drug are the most important factors affecting the pharmacokinetics of drugs. Drug doses used in these patients are recommended to be calculated according to total body weight (TVA), ideal body weight (IVA), and lean body weight (HVA = IVA + 20%), taking into account the lipophilic nature of the drug. For example in induction; when using high lipophilic drugs according to YVA or IVA; moderately lipophilic For drugs, the dosage can be increased by 20-40% and used according to the YVA.Propofol's high lipophilic properties cause its effect to start very quickly and to be short-lived. It has been shown in many studies that there is no usable accumulation or prolongation of propofol compared to TVA in obese patients.

Short-acting remifentanil, one of the lipophilic synthetic opioids, can be administered according to IVA .

There are no well-known guidelines for intraoperative fluid management in bariatric surgery. Different intraoperative fluid management protocols are used. The key to improving outcomes from treatment in the post-operative period is "patient directed fluid management" or "targeted fluid management". The use of Perioperative Goal-Directed Fluid Therapy Technologies helps the anesthesiologist to closely monitor the patient and establish the delicate balance between benefit and risk. Plethysmographic variability index monitoring (PVI-Pleth Variability Index) is a non-invasive, automatic and continuous monitor that displays the fluid response of patients, and is one of the easy-to-apply and easily interpreted monitoring methods. It has been shown that intraoperative hypotension and fluid need can be predicted with PVI monitoring.

The aim of this study is to determine the effect of Pleth Variability Index (PVI) monitoring on intraoperative volume replacement amount and postoperative complications in obese patients who underwent bariatric surgery.

Patients and Methods

Patients A total of 60 obese patients who scheduled for elective bariatric surgery were included in this single-blind prospective randomized study. Patients were required to have an ASA physical status class 2 or 3. Exclusion criteria were as follows: severe cardiac arrhythmia, peripheral artery disease, an ejection fraction <30%, any pulmonary pathology preventing a respiratory volume >6 ml/kg/min on mechanical ventilation, and hepatic or renal impairment. The study protocol was approved by the local ethics committee of Marmara University Medical Faculty (03.01.2020- 09.2020.158). All patients provided informed consent prior to study entry and the study was conducted in accordance with the Declaration of Helsinki.

Study groups Patients were randomly assigned to the PVI group or control group using sealed envelope method. Fluid management was based on PVI values in the PVI group, where a PVI value <13% was targeted throughout the operation. Standard fluid management regimen was used for the controls. All patients fasted for eight hours before the operation. In the operating room, all patients were monitored for PVI; however, anesthesia team was able to see only the PVI values of the PVI groups that would aid fluid management; whereas team was blinded to the PVI values of the controls in whom the fluid management was done using standard approach. On the other hand, PVI values of the controls were also recorded by another anesthesiologist every 15 minutes.

Anesthesia management For anesthesia induction, 2 mg/kg propofol and 1μgr/kg remifentanil were used in all patients and 0.6 mg/kg rocuronium (Esmeron vial, Schering -Plough, Istanbul, Turkey) was used for muscle relaxation. Following endotracheal intubation, total intravenous anesthesia with propofol and remifentanil was used. In addition to PVI, both groups were monitored for other parameters such as heart rate (HR), noninvasive mean blood pressure (MAB), and perfusion index (PI), and bispectral index scale (BIS). Propofol dose was adjusted to keep BIS between 40 and 45 throughout the operation.

Fluid management Controls Following anesthesia induction, controls received crystalloid solution at an infusion rate of 4-8 ml/kg/h for fluid maintenance. Infusion rate was adjusted by the same anesthesiologist based on routine approach based on intraoperative assessments such as heart rate, mean arterial pressure and urine output. In case of hypotension, which was defined as mean arterial blood pressure <65 mmHg, crystalloid infusion was increased and colloid infusion (Gelofusine® Melsungen, Germany) was started. In case hypotension persists, 5 mg of ephedrine was administered intravenously, and it was repeated every 5 minutes until mean arterial blood pressure is above 65 mmHg.

PVI group Crystalloid replacement was adjusted according the PVI values, which were targeted to be kept below 13% above 5%. Fluid maintenance was started with 2ml/kg/hour crystalloid dose. If PVI is >13% for more than 5 minutes, a 250 ml bolus Gelofusine® was administered. If PVI was still >13% following this, it was repeated every 5 minutes until PVI<13%. Meanwhile, 5 mg bolus ephedrine was administered to keep mean blood pressure over 65 mmHg, when necessary. In case mean blood pressure is <65 mmHg, intravenous 5 mg ephedrine was repeated every 5 minutes until mean blood pressure is over 65 mmHg.

Assessments Following parameters were recorded intraoperatively at 15 minutes intervals: PVI value, heart rate, mean arterial pressure, perfusion index value. In addition, preoperative bun, creatinine, and lactate values, perioperative use of crystalloids, colloids, blood/blood products, and bleeding amounts, intra- and postoperative urine outputs, as well as postoperative bun, creatinine, lactate values were recorded.

ELIGIBILITY:
Inclusion Criteria:

* obese patients who scheduled for elective bariatric surgery

Exclusion Criteria:

* severe cardiac arrhythmia
* peripheral artery disease
* an ejection fraction <30%
* any pulmonary pathology preventing a respiratory volume >6 ml/kg/min on mechanical ventilation
* hepatic or renal impairment

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: sample size 60
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Fluid therapy in bariatric patients | during surgery
  Fluid therapy is providewith pleth variability index monitorisation

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)